CLINICAL TRIAL: NCT04850703
Title: Comparative Study of the Clinical Response Between tDCS and Dapoxetine, Define a Very Effective Therapeutic Target, That Improves the LPE in the Medium Long Term
Brief Title: Brain Networks Implicated in Lifelong Premature Ejaculation Patients
Acronym: LPE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Moises Domingo (Other)
Collaborators: Dr. Alejandro Molina Cabeza (Unknown); Susana Ferrandis Martinez (Unknown)
Responsible Party: Sponsor-Investigator, Moises Domingo, Sub Investigator, Spanish Foundation for Neurometrics Development
Organization: Spanish Foundation for Neurometrics Development (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0104201UR
Record Dates: First submitted 2021-04-07; First posted 2021-04-20 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Premature Ejaculation; Sexual Dysfunction
Keywords: Brain Mapping; EEG; ERP; tDCS; tRNS; Dapoxetine; Lifelong premature ejaculation; central inhibitory network function; inferior frontal gyrus; dentate nucleus; right frontal pole; Resting State Networks; Funtional connectivity
MeSH Terms: conditions — Premature Ejaculation; Sexual Dysfunction, Physiological

STUDY DESIGN:
Intervention Model Description: Allocation: Randomized Intervention Model: Parallel Assignment
Who Masked: Care Provider, Investigator
Masking Description: 12 patients will be receive tRNS sham 10 sessions. 12 patients will take Dapoxetine, sham 10.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Premature Ejaculation participants who receive Brain Weak Currents in IFG brain cortex (Experimental): Participants receive tRNS (weak currents < 2 mA) sessions at IFG brain cortex for 25 minutes 2 times a day 3 times per week during 3 weeks.
  After 4 hours they end the last session, a new brain mapping is performed.
  Interventions: Device: Transcranial Radom Noise Stimulation
- Premature Ejaculation participants who take Dapoxetine (Active Comparator): Participants take 1 tablet of the drug between 1 and 3 hours before the brain mapping
  Interventions: Drug: Take Dapoxetine
- Placebo Group (Sham Comparator): Participants who do not take medication or receive tRNS sessions
  Interventions: Combination Product: Comparation EEG changes between Sham Group against tRNS and Dapoxetin participants
- Controls (Other): 44 Healthy humans not clinically not diagnosed with LPD and withouth expression the LPE endophenotype. In this way, the investigators what would be the patients diagnosed clinically with LPE who present the endophenotype or neurophysiological biomarker of LPE.
  Interventions: Diagnostic Test: Compare LPE EEG endophenotype between participants and healthy controls

INTERVENTIONS:
Device: Transcranial Radom Noise Stimulation — tRNS against Dapoxetine in LPE patients
  Other Names: tRNS
  Arms: Premature Ejaculation participants who receive Brain Weak Currents in IFG brain cortex
Drug: Take Dapoxetine — Dapoxetine against tRNS in LPE patients
  Arms: Premature Ejaculation participants who take Dapoxetine
Combination Product: Comparation EEG changes between Sham Group against tRNS and Dapoxetin participants — Compare EEG parameters like Theta Rhythm and Coherence between three groups of participants: sham, tRNS participants and Dapoxetine participants groups.
  Arms: Placebo Group
Diagnostic Test: Compare LPE EEG endophenotype between participants and healthy controls — Define as precisely as possible the electrophysiological endophenotype of Longlife Premature Ejaculation, using healthy humans who do not express the LPE EEG endophenotype
  Arms: Controls

SUMMARY:
Using Brain Mapping and Cognitive ERPs, the investigatos have searched for a Brain Networks involved during Inhibitory Control in Lifelong Premature Ejaculation (LPE) participants. The investigators have designed a clinical trial comparing placebo with tDCS and blacebo group against Dapoxetine, studying the effects on LPE, as well as side effects and their medium and long-term duration.

DETAILED DESCRIPTION:
Lifelong premature ejaculation (LPE) is a very common male sexual dysfunction like erectile dysfunction. It produces great distress to sexual harmony and even fertility. Previous neurophysiology studies revealed an ejaculation-related control mechanism in the brain: left inferior frontal gyrus (IFG) activation during successful inhibition. If we use the left IFG as a seed, participants showed weaker resting-state functional connectivity (FC) activity, between the seed and two areas (left dentate nucleus (DN) and right frontal pole) compared with controls.

The main goal is to compare whether the brain biomarker only exists in participants with LPD and how it responds to treatment with Dapoxetine and with tDCS against the IFG networks and lDN, measuring the connectivity changes in these brain networks and FC.

ELIGIBILITY:
Inclusion Criteria:

* To be over 18 years old and less than 70 years
* Best-practice diagnosed Longlife Premature ejaculation
* Diagnosed since at least one years prior to enrollment.
* No use drugs or medicines

Exclusion Criteria:

* Serious visual and hearing loss
* Brain injury following cranial trauma
* Other neurological disorders like Parkinson, ME, headache, etc.
* Birth trauma
* Mental retardation

Ages: 30 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — All of patients were diagnosed of Longlife Premature Ejaculation
Enrollment: 128 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2022-05-21 (Actual); Study Completion 2023-02-04 (Actual)

PRIMARY OUTCOMES:
Wavelet Changes define Brain Biomarker of LPE | 1 month
  The investigators will reported changes in wavelet (time-frequencies) in Left Prefrontal Lobe F3, F7 and Fz electrodes.
EEG coherence comparing Dapoxetine against tRNS | 2-3 months
  The investigators will reported changes in brain connectivity comparing taking Dapoxetine with the use of tRNS, calculating EEG coherence.
Adverse events comparing Dapoxetine against tRNS | 2-3 months
  Report adverse events during the application of the protocol Dapoxetine / tRNS.

SECONDARY OUTCOMES:
Measure the effect of Dapoxetine through ERP Novelty Wave comparing with the values of the controls | 1 month
  Changes in latencies and amplitude of Novelty wave in the Ventro-lateral prefrontal cortex comparing novelty wave in Dapoxetine group against controls.
Measure the effect of tRNS through ERP Novelty Wave changes comparing with the values of the controls | 1 month
  Changes in latencies and amplitude of Novelty wave in the Ventro-lateral prefrontal cortex comparing novelty wave in tRNS group against controls.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Molina Cabeza, MD, Principal Investigator — Sexual Salud Valclinic
Locations (1):
- Salud Valclinic, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sexual Valclinic health Institute — https://saludsexualvalclinic.com/
- See also: Urology Department Hereford Hospital — http://herefordshireurology.co.uk/